CLINICAL TRIAL: NCT01831869
Title: The Beneficial Effect of L-Thyroxine Long -Term Replacement on Lipid Profiles and Atherosclerosis in Subclinical Hypothyroidism: A Prospective Study
Brief Title: Effect of L-Thyroxine on Lipid Profiles and Atherosclerosis in Subclinical Hypothyroidism
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Ling Gao, Professor, Shandong Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012GSF11824
Record Dates: First submitted 2013-04-07; First posted 2013-04-15 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Hypothyroidism; Thyroid Diseases; Endocrine System Diseases
Keywords: Subclinical hypothyroidism; L-thyroxine; Lipid; endothelial function; inflammatory factor; adipocytokine
MeSH Terms: conditions — Hypothyroidism; Thyroid Diseases; Endocrine System Diseases | interventions — Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L-thyroxine (Active Comparator): Oral administration, starting dose 25 or 50 micrograms once daily.
  Interventions: Drug: L-thyroxine
- blank (No Intervention): no intervention

INTERVENTIONS:
Drug: L-thyroxine
  Arms: L-thyroxine

SUMMARY:
Subclinical hypothyroidism (SCH) is a common condition affecting 3-10% of the general population, especially in women older than 50 years old. It is controversial whether SCH can lead to increased risks of cardiovascular (CV) disease and whether treatment with L-thyroxine reverses these risks. The present study was designed to evaluate the effect of L-thyroxine treatment in SCH on lipid profile, atherosclerosis, endothelial function, serum inflammatory factors and adipocytokines.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged of 18 to 60 years old;
* Diagnosis was subclinical hypothyroidism(elevated serum thyroid-stimulating hormone levels with normal serum free T4 levels measured at least two times with a three-month interval);
* untreated.

Exclusion Criteria:

* Pregnancy or lactation women;
* Presence of pituitary/hypothalamic disorders, diabetes mellitus or other endocrinal and metabolic disorders;
* Presence of psychological or physical disabilities,acute infection, cerebrovascular or cardiovascular disease, chronic respiratory disease and other illnesses known to alter lipid metabolism;
* Taking lipid-lowering agents and other drugs that known to influence thyroid function, blood pressure, heart function or bile acids;
* Obviously poor compliance.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2013-04; Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
change in lipid profile | measured at baseline; 6 month; 12 months and 24 months.
change in thickness of blood vessel wall | measured at baseline; 6 months; 12 months and 24 months.

SECONDARY OUTCOMES:
change in endothelial function | measured at baseline; 6 months; 12 months and 24 months.
change of adipocytokines | measured at baseline; 6 months; 12 months and 24 months.
Change of Oxidative Stress and Chronic Inflammatory Factors Related with Atherosclerosis | measured at baseline; 6 months; 12 months and 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jiajun Zhao, Study Chair — Shandong Provincial Hospital
Locations (1):
- Shandong Provincial Hospital, Jinan, Shandong, China